CLINICAL TRIAL: NCT03599466
Title: Clinical Bioequivalence Study on Two Lisinopril Tablets 20mg Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited (Industry)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BABE-P15-099
Record Dates: First submitted 2018-01-16; First posted 2018-07-26 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — Lisinopril

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BF-Lisinopril Tablets 20mg (Experimental): During the study session, the subjects will be administered a single dose of BF-Lisinopril Tablet 20mg after an overnight fast of approximately 10 hours.
  Interventions: Drug: BF-Lisinopril Tablets 20mg; Drug: Zestril Tab 20mg
- Zestril Tab 20mg (Active Comparator): During the study session, the subjects will be administered a single dose of Zestril Tab 20mg after an overnight fast of approximately 10 hours.
  Interventions: Drug: BF-Lisinopril Tablets 20mg; Drug: Zestril Tab 20mg

INTERVENTIONS:
Drug: BF-Lisinopril Tablets 20mg — BF-Lisinopril Tablets 20mg is a generic product manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited
Drug: Zestril Tab 20mg — Zestril Tab 20mg will be used as a reference drug in this study

SUMMARY:
The objective of the study is to compare the bioavailability of a generic product of lisinopril with that of a reference product when administered to healthy volunteers under fasting condition. The test product is BF-Lisinopril Tablet 20mg (HK-63564) manufactured by Bright Future Pharmaceuticals Factory O/B Bright Future Pharmaceutical Laboratories Limited, and the reference product is Zestril Tab 20mg (HK-30515). The bioequivalence or bioinequivalence of the test and reference formulations will be assessed and concluded based on the plasma pharmacokinetic data of lisinopril, as well as WHO guidelines on registration requirements to establish interchangeability.

DETAILED DESCRIPTION:
It is planned to enroll 16 to 30 healthy subjects, with an aim to obtain at least 12 evaluable subjects. The study design is a single-dose, two-treatment, two-period, two-sequence crossover with a washout period of one to two weeks. During each study session, the subjects will be administered a single dose of 20mg lisinopril (one BF-Lisinopril tablets 20mg or one Zestril Tab 20mg) after an overnight fast of approximately 10 hours. Venous blood samples will be collected at pre-dose (0h) and at 1,2,4,5,6,7,8,9,10,12,24 and 48 hours post-dose (13 time points). The plasma concentrations of lisinopril will be determined by a validated assay. The non-compartmental method will be used to analyze the plasma concentration-time data and calculate the main pharmacokinetic parameters such as Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. ANOVA will be calculated on logarithmically transformed Cmax, AUC0-last and AUC0-inf. The two one sided tests will be used to calculate the 90% confidence intervals for the mean difference in AUC0-last, AUC0-inf and Cmax and to assess the bioequivalence of the two products.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female, 18 to 55 years of age
* Body Mass Index between 18 to 30 kg/m2
* Accessible vein for blood sampling
* High probability for compliance and completion of the study
* Female subjects must agree to practice abstinence or take effective contraceptive methods to prevent pregnancy from the start of the screening and until two weeks of last dose administration.

Exclusion Criteria:

* Clinically significant hepatic, renal, biliary, cardiovascular, gastrointestinal, haematological and other chronic and acute diseases within 3 months prior to the study
* Clinically significant abnormality in physical examination, vital sign, laboratory test results, ECG evaluation, urine test, blood chemistry or haematological test
* Regular consumption of tobacco used in any forms
* Regular consumer of alcohol (more than one drink per day)
* Blood donation within 4 weeks prior to the start of the study
* Use of lisinopril within 4 weeks before the study
* Use of antihypertensive medications or angiotensin-converting enzyme (ACE) inhibitors within 4 weeks before the study
* Volunteer in any other clinical drug study within 2 months prior to this study
* Hypersensitivity to lisinopril or other drugs in its class
* History of drug abuse in any form
* Female subjects who are breastfeeding or pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of Lisinopril | 48 hours
  Peak drug concentration, obtained directly from the original concentration-time data.
Area under the plasma concentration versus time curve (AUC) of Lisinopril | 48 hours
  Area under the concentration-time curve from time zero to the last sampling time.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) of Lisinopril | 48 hours
  Time to peak drug concentration, obtained directly from the original concentration-time data.
Elimination half-life (t1/2) of Lisinopril | 48 hours
  Terminal elimination half-life, calculated as 0.693/(the terminal phase elimination rate constant that can be obtained using WinNonlin)

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Zuo, Principal Investigator — School of Pharmacy, The Chinese University of Hong Kong; Riza Ozaki, Study Director — Phase 1 Clinical Trial Centre, The Chinese University of Hong Kong; Brian Tomlinsion, Study Director — Department of Medicine and Therapeutics, The Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Study investigators and his/her study team members, domestic and foreign regulatory agencies, members of ethics committee and health authorities, monitors and auditors relevant to conduct of this clinical study will be granted free access to subject's data. The relevant technical, medical, pharmaceutical, biological and chemical personnel of the sponsor will have access to the case report forms.